CLINICAL TRIAL: NCT00473642
Title: A Prospective Pilot Study of Reduced Fluence Photodynamic Therapy With Visudyne® (Verteporfin) in Combination With Lucentis™ (Ranibizumab) for the Treatment of Age-Related Macular Degeneration
Brief Title: Reduced Fluence Photodynamic Therapy (PDT) With Visudyne in Combination With Lucentis for Age-Related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007002
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Age-Related Maculopathy; Choroidal Neovascularization
Keywords: Ranibizumab; Lucentis; Verteporfin; Visudyne; Photodynamic therapy
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Standard Fluence Photodynamic Therapy combined with ranibizumab
  Interventions: Drug: Ranibizumab; Drug: Verteporfin
- 2 (Experimental): Verteporfin at 50% fluence photodynamic therapy combined with ranibizumab
  Interventions: Drug: Ranibizumab; Drug: Verteporfin
- 3 (Active Comparator): Ranibizumab monotherapy
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — intravitreal administered ranibizumab 0.5 mg in 0.05 mL
  Other Names: Lucentis
Drug: Verteporfin — Verteporfin with 50% fluence photodynamic therapy (25 J/cm2)
  Other Names: Visudyne
  Arms: 2
Drug: Verteporfin — Verteporfin with standard fluence photodynamic therapy (50 J/cm2)
  Other Names: Visudyne
  Arms: 1

SUMMARY:
In this pilot study the researchers will evaluate the safety and efficacy of 50% reduced fluence PDT combination therapy with ranibizumab. The researchers hope to gain information regarding the use of reduced fluence PDT combination therapy. The information gained from this pilot study may prompt further definitive studies comparing the safety and efficacy of both standard fluence PDT combination therapy, reduced fluence PDT combination therapy, and ranibizumab monotherapy.

The study will compare the use of combination therapy with ranibizumab and verteporfin PDT to ranibizumab alone in patients with exudative age-related macular degeneration (AMD). All patients will receive three consecutive monthly treatments with ranibizumab. Patients will be randomized 1:1:1 to 3 groups. Patients randomized to group 1 will receive only ranibizumab. Patients randomized to group 2 will also receive one treatment with reduced fluence (50% fluence) verteporfin PDT at day 0. Patients randomized to group 3 will also receive one treatment with standard fluence verteporfin PDT. All patients will also be evaluated for possible retreatment with ranibizumab and verteporfin PDT according to established criteria. Thirty patients will be recruited from one U.S. sites. Randomization will occur at the time of entry into the study. Follow-up will continue until month 12 (from day 0) in all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female Patients > 50 years of age.
2. Patients with primary subfoveal CNV secondary to AMD documented on IVFA and/or OCT.
3. Patient with BCVA of 20/40 to 20/320 in the study eye using Early Treatment Diabetic Retinopathy Study (ETDRS) charts. See definition of ETDRS charts.
4. If both eyes are eligible, only one eye will be evaluated in the study. The eye with lesser visual acuity will be selected as the study eye.
5. Patients must be able and willing to provide written informed consent.

Exclusion Criteria:

1. Patients receiving prior treatment in the study eye with verteporfin, any focal laser photocoagulation, vitrectomy, or intravitreous injection of antiangiogenic medications, including triamcinolone, pegaptanib, bevacizumab, or ranibizumab.
2. Neovascular membrane from any other retinal disease such as myopic degeneration, histoplasmosis, retinal angiomatous proliferation, or other ocular inflammatory disease.
3. Choroidal neovascular membrane greater than 9 disc diameters in size.
4. Previous posterior vitrectomy in the study eye.
5. Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period.
6. Pregnant women or premenopausal women not using adequate contraception.
7. History of allergy to fluorescein, Visudyne, Lucentis.
8. Inability to comply with study or follow up procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Westhouse, DO, Principal Investigator — Oklahoma State University Medical Center; Raymond Townsend, MD, Principal Investigator — Oklahoma State University Medical Center; John Saurino, DO, Principal Investigator — Oklahoma State University Medical Center
Locations (1):
- Eagle Mountain Vision, Tulsa, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Fluence PDT: Standard Fluence Photodynamic Therapy combined with ranibizumab
- 50% Fluence PDT: Verteporfin at 50% fluence photodynamic therapy combined with ranibizumab
- Ranibizumab: Ranibizumab monotherapy
Period: Overall Study
Arm/Group | Standard Fluence PDT | 50% Fluence PDT | Ranibizumab
Started | 10 | 11 | 10
Completed | 8 | 10 | 8
Not Completed | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Fluence PDT | 50% Fluence PDT | Ranibizumab | Total
Number analyzed (Participants) | 10 | 11 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 4
  >=65 years | 9 | 9 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (3.1) | 73.4 (2.1) | 76.3 (2.8) | 74 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 23
  Male | 2 | 4 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in BCVA of ETDRS Letters From Baseline at 12 Months
Description: Visual acuity is often measured using a chart called the ETDRS chart (Early Treatment Diabetic Retinopathy Study). A letter score is calculated based on the number of letters that can be correctly identified from specified distances. Higher letter scores correspond to better visual acuity. Lower letter scores mean poorer visual acuity. In this study the baseline visual acuity in letters is subtracted from the visual acuity in letters measured at the 12 month visit providing a letter score of vision gain or vision loss.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Letters
Groups:
- Standard Fluence PDT: Standard Fluence Photodynamic Therapy combined with ranibizumab
  Ranibizumab: intravitreal administered ranibizumab 0.5 mg in 0.05 mL
  Verteporfin: Verteporfin with standard fluence photodynamic therapy (50 J/cm2)
- Reduced Fluence PDT: Verteporfin at 50% fluence photodynamic therapy combined with ranibizumab
  Ranibizumab: intravitreal administered ranibizumab 0.5 mg in 0.05 mL
  Verteporfin: Verteporfin with 50% fluence photodynamic therapy (25 J/cm2)
- Ranibizumab Monotherapy: Ranibizumab monotherapy
  Ranibizumab: intravitreal administered ranibizumab 0.5 mg in 0.05 mL
Arm/Group | Standard Fluence PDT | Reduced Fluence PDT | Ranibizumab Monotherapy
Number analyzed (Participants) | 10 | 11 | 10
Letters | 5.9 [-0.4 to 12.2] | 7.6 [3.6 to 11.6] | 16.4 [12.4 to 20.4]

2. Primary Outcome: Mean Letters Gained of Best Corrected Visual Acuity Using ETDRS Protocol
Description: as for outcome 1
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Standard Fluence PDT | 50% Fluence PDT | Ranibizumab
Number analyzed (Participants) | 10 | 11 | 10
letters | 5.9 (6.3) | 7.6 (4) | 16.4 (4)

3. Secondary Outcome: Time to First Retreatment After Loading Doses
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Month
Arm/Group | Standard Fluence PDT | Reduced Fluence PDT | Ranibizumab Monotherapy
Number analyzed (Participants) | 10 | 11 | 10
Month | 2.86 (0.38) | 2.90 (0.71) | 2.86 (0.63)

4. Secondary Outcome: Average Number of PDT Retreatments Over 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Treatments
Arm/Group | Standard Fluence PDT | Reduced Fluence PDT
Number analyzed (Participants) | 10 | 11
Number of Treatments | 0.67 (0.24) | 0.55 (0.22)

5. Secondary Outcome: Central Macular Thickness Reduction on OCT
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: micron (um)
Arm/Group | Standard Fluence PDT | Reduced Fluence PDT | Ranibizumab Monotherapy
Number analyzed (Participants) | 10 | 11 | 10
micron (um) | 42.9 (20.1) | 76.1 (37.8) | 34.9 (10.9)

6. Secondary Outcome: Average Number of Ranibizumab Retreatments Over 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Treatments
Arm/Group | Standard Fluence PDT | Reduced Fluence PDT | Ranibizumab Monotherapy
Number analyzed (Participants) | 10 | 11 | 10
Number of Treatments | 2.67 (0.53) | 2.91 (0.62) | 4.14 (0.72)

ADVERSE EVENTS:
Arm/Group | Standard Fluence PDT | 50% Fluence PDT | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 2/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Fluence PDT (N=10) | 50% Fluence PDT (N=11) | Ranibizumab (N=10)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — greater than 2 months after last ranibizumab
cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — following hip fracture and complications greater than 2 months after ranibizumab

LIMITATIONS AND CAVEATS:
This study was limited by a small number of subjects. Additionally, several subjects did not meet the 12 month study endpoint. These subjects were included in the final analysis if their last visit was within 2 months of the final endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less